CLINICAL TRIAL: NCT03861715
Title: Single Follicular Dexarelix, a New Long Acting GnRH- Antagonist for LH Suppression During Ovarian Stimulation in Oocyte Donors. A Randomised Control Trial.
Brief Title: Single Follicular Dexarelix for LH Suppression During Ovarian Stimulation in Oocyte Donors.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assisting Nature (Other)
Responsible Party: Principal Investigator, Papanikolaou Evaggelos, Papanikolaou Evaggelos, MD, PhD, Fertility Specialist, Scientific Director at Assisting Nature IVF Clinic, Assisting Nature
Other Study IDs: Single-VS-multiple dose- AN007
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Infertility; Premature Ovarian Failure
Keywords: antagonist protocol; degarelix antagonist protocol; degarelix; IVF
MeSH Terms: conditions — Infertility; Primary Ovarian Insufficiency | interventions — Pregnancy Rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Single Dose antagonist Degarelix: The blastocyst formation rate and live birth rates of patients who followed GnRH antagonist protocol with a single dose Degarelix.
  Interventions: Diagnostic Test: live birth rate
- Multidose antagonist Ganirelix: The blastocyst formation rate and live birth rates of patients who followed GnRH antagonist protocol with multidose dose Ganirelix.
  Interventions: Diagnostic Test: live birth rate

INTERVENTIONS:
Diagnostic Test: live birth rate — The blastulation rate and live birth rate according to the protocol of COS
  Other Names: blastulation rate

SUMMARY:
A randomized prospective study in the evaluation of the long acting GnRH antagonist Degarelix against the classical multidose regime with Ganirelix for LH suppression during the follicular phase of an ovarian stimulation cycle in oocyte donors.

DETAILED DESCRIPTION:
A randomized prospective study of the use of single dose of the long acting GnRH antagonist Degarelix for ovarian stimulation cycle in oocyte donors: Ovarian stimulation started on cycle Day2 with gonadotropins 175-300 IU and either GnRH antagonist single dose Degarelix or multidose GnRH antagonist Ganirelix initiated on Day6 of the stimulation cycle. Agonist triggering was used in both groups for oocyte maturation. Blastocyst formation rate and Live Birth Rates were estimated for both groups.

ELIGIBILITY:
Inclusion Criteria:

* age 20-34 years;
* body mass index (BMI) 18-29kg/m2;
* regular menstrual cycle of 26-35 days,
* AMH levels age appropriate (≥2.3 ng/ml)
* early follicular- phase serum concentration of FSH within normal limits (1-12 IU/l).

Exclusion Criteria:

* women with diabetes and other metabolic disease
* women with hereditary genetic diseases;
* women with heart disease, QT prolongation,heart failure
* elevated liver enzymes, liver failure, hepatitis
* women with inflammatory or autoimmune disease
* abnormal karyotype;
* endometriosis stage III/IV;
* history of recurrent miscarriage;
* severe OHSS in a previous stimulation cycle or any contraindication for the use of gonadotrophins.

Ages: 20 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women 20-34 years old who follow COS with a single GnRH antagonist Degarelix or multidose GnRH antagonist Ganirelix.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Live birth rate according to stimulation protocol | Up to 38 weeks after embryo transfer
  Live birth rate according to stimulation protocol

SECONDARY OUTCOMES:
Blastulation rate according to stimulation protocol | Up to 6 days post oocyte retrieval
  Blastulation rate according to stimulation protocol

CONTACTS AND LOCATIONS:
Overall Officials: Evaggelos Papanikolaou, MD, PhD, Principal Investigator — Assisting Nature; Robert Najdecki, MD, PhD, Principal Investigator — Assisting Nature
Locations (1):
- Assisting Nature, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: Undecided